CLINICAL TRIAL: NCT03314155
Title: Cerebral Neuroinflammation During Major Depressive Episode: Multicentric Comparative Study.
Brief Title: Cerebral Neuroinflammation During Major Depressive Episode
Acronym: InflaDep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/16/8918; 2017-001478-40 (EudraCT Number)
Record Dates: First submitted 2017-08-21; First posted 2017-10-19 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Depressive Disorder
Keywords: Depressive disorder; Treatment Resistant Depression; [18 F ] DPA- 714; PET; MRI; Inflammation
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Treatment-Resistant; Inflammation

STUDY DESIGN:
Masking Description: Images' analysis will be done by an INSERM engineer without the knowledge of the group to which the subjects belong.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cerebral neuroinflammation evaluation (Experimental): The density of TSPO (which is an inflammation maker) is evaluated by the tracer's brain distribution volume ([18F] DPA-714).
  Interventions: Diagnostic Test: Cerebral neuroinflammation evaluation

INTERVENTIONS:
Diagnostic Test: Cerebral neuroinflammation evaluation — Pet scan following an injection of the radiotracer ([18F]DPA-714), to evaluate the neuroinflammation. MRI to evaluate functional and structural integrities. Blood test to analyze various inflammation marker (IL-6, Tumor Necrosis Factor (TNF) alpha, CRPus, and TSPO). And psychological scales to assess the depressive symptoms.

SUMMARY:
the investigators make the following assumptions: 1) neuroinflammation in MDD can be measured by the [18 F ] DPA- 714 ; 2) it is accompanied by anatomical and functional changes in the frontal subcortical loops, strongly involved in MDD ; 3) neuroinflammation in patients might be a biomarker related to resistance to treatment in patients with MDD. If this assumptions are validated, then this study will enable a better understanding of the neuroinflammatory processes. This breakthrough could have a long term therapeutic impact, helping to target more specifically antidepressant drugs with anti-inflammatory action and / or drugs targeting neuroinflammation.

DETAILED DESCRIPTION:
The most widespread pathophysiological hypothesis in major depressive disorder (MDD), is the hypothesis of monoamine deficit. The most used antidepressants in everyday clinical practice act by inhibiting the reuptake of monoamines. However, meta-analyzes evaluating the efficacy of antidepressants suggest that they are ineffective in 30 to 40% of patients. Inflammatory mechanisms might be related to the deficiency of monoamines, compromising the effectiveness of conventional antidepressants. Newly developed specific radiotracers allow the use of positron emission tomography (PET) imaging techniques to evaluate neuroinflammation. It has recently demonstrated the relevance of the [18F] DPA- 714 as a biomarker of neuroinflammation in humans in several neurological diseases.

ELIGIBILITY:
* Inclusion criteria for all groups:

  * Written agreement for participation
  * Able to understand instructions and information data
* Inclusion criteria for the experimental group:

  * Responding to MDD criteria (DSM-5)
  * MADRS score> 20
  * Antidepressant medication considered ineffective and before the introduction of a new treatment according to the recommendations (unchanged dosage for at least a week and plasma levels within the therapeutic range)
* Inclusion criteria for the pathological control group :

  * Having met MDD criteria (DSM-5)
  * In remission for 8 weeks according to the DSM-5
  * MADRS score <10
  * Treated with antidepressants (unchanged dosage for at least week)
* Inclusion criteria for the control group :

  * Without any neurological or psychiatric previous disorder
  * CRPus < 5mg/L
* Exclusion criteria for all groups:

  * Patients without public insurance regime.
  * Specific contraindication to the use of MRI (metallic material) or PET (specific allergy related to the ligand).
  * Pregnant and breastfeeding women
  * Persons deprived of liberty by judicial or administrative decision
  * People hospitalized without consent, or subject to legal protection
  * Persons unable to consent
  * Patients with a neurodegenerative disease, bipolar disease, chronic psychotic disorder, addictive disorder, Obsessive Compulsive Disorder, Post-Traumatic Stress disorder (PCL-S> ou =45), known system pathology
  * Patients with a history of stroke
  * Patients with an acute infectious disease
  * Patients with chronic inflammatory pathology.
  * Patients treated with anti-inflammatory and/or immunosuppressive, and/or antipsychotics, and/or diazepam
* Exclusion criteria for control group:

  * No significant psychiatric or somatic history.
  * No psychotropic treatment
  * Suicidal risk (C-SSRS)
  * Anxiety Disorders (MINI)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
distribution pattern of neuroinflammation in Positron Emission Tomography (PET) data | Day 7
  Assessed between patients with MDD (experimental group), patients who have had a MDD and being in remission for at least 8 weeks, still treated with antidepressants, matched in age and gender with the experimental group (pathological control group) and control subjects, matched in gender and age with both patients' groups (control group).

SECONDARY OUTCOMES:
distribution pattern of neuroinflammation in PET data across all groups | Day 7
  Across all groups (i.e. experimental group, pathological control group and control group).
patients with depressive symptoms and neuroinflammation (i.e. PET data). | Day 7
  Depressive symptoms are assessed by the Montgomery and Asberg Depression Scale (MADRS) and the Columbia-Suicide severity rating scale (CSSRS).
  Correlation across all groups (experimental group, pathological control group and control group).
patients with neuroinflammation (i.e. PET analysis) and MRI parameters for functional and structural integrities. | Day 7
  Correlation across all groups (experimental group, pathological control group and control group).
patients with neuroinflammation (i.e. PET analysis) and biological markers of neuroinflammation (i.e. cytokines). | Day 7
  Correlation across all groups (experimental group, pathological control group and control group).

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Yrondi, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - Hôpital de Psychiatrie, Toulouse, Midi-Pyrénées
  - CHU Bordeaux, Bordeaux, Nouvelle-Aquitaine
  - CHRU Lapeyronie, Montpellier, Occitanie
  - Clinique Psychiatrique Universitaire CHRU Tours, Tours, Val-De-Loire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sartorius N. The economic and social burden of depression. J Clin Psychiatry. 2001;62 Suppl 15:8-11. PMID 11444765
- [Background] Bakish D. New standard of depression treatment: remission and full recovery. J Clin Psychiatry. 2001;62 Suppl 26:5-9. PMID 11775091
- [Background] Papakostas GI, Petersen T, Mahal Y, Mischoulon D, Nierenberg AA, Fava M. Quality of life assessments in major depressive disorder: a review of the literature. Gen Hosp Psychiatry. 2004 Jan-Feb;26(1):13-7. doi: 10.1016/j.genhosppsych.2003.07.004. PMID 14757297
- [Background] Schildkraut JJ, Schanberg SM, Breese GR, Kopin IJ. Norepinephrine metabolism and drugs used in the affective disorders: a possible mechanism of action. Am J Psychiatry. 1967 Nov;124(5):600-8. doi: 10.1176/ajp.124.5.600. No abstract available. PMID 4383104
- [Background] Maes M, Noto C, Brietzke E. Omics-based depression and inflammation research. Braz J Psychiatry. 2015 Jan-Mar;37(1):1-2. doi: 10.1590/1516-4446-2015-3609. No abstract available. PMID 25806550
- [Background] Hasler G, van der Veen JW, Tumonis T, Meyers N, Shen J, Drevets WC. Reduced prefrontal glutamate/glutamine and gamma-aminobutyric acid levels in major depression determined using proton magnetic resonance spectroscopy. Arch Gen Psychiatry. 2007 Feb;64(2):193-200. doi: 10.1001/archpsyc.64.2.193. PMID 17283286
- [Background] Deschwanden A, Karolewicz B, Feyissa AM, Treyer V, Ametamey SM, Johayem A, Burger C, Auberson YP, Sovago J, Stockmeier CA, Buck A, Hasler G. Reduced metabotropic glutamate receptor 5 density in major depression determined by [(11)C]ABP688 PET and postmortem study. Am J Psychiatry. 2011 Jul;168(7):727-34. doi: 10.1176/appi.ajp.2011.09111607. Epub 2011 Apr 15. PMID 21498461
- [Background] Entsuah AR, Huang H, Thase ME. Response and remission rates in different subpopulations with major depressive disorder administered venlafaxine, selective serotonin reuptake inhibitors, or placebo. J Clin Psychiatry. 2001 Nov;62(11):869-77. doi: 10.4088/jcp.v62n1106. PMID 11775046
- [Background] Blumberg HP, Kaufman J, Martin A, Whiteman R, Zhang JH, Gore JC, Charney DS, Krystal JH, Peterson BS. Amygdala and hippocampal volumes in adolescents and adults with bipolar disorder. Arch Gen Psychiatry. 2003 Dec;60(12):1201-8. doi: 10.1001/archpsyc.60.12.1201. PMID 14662552
- [Background] Stone VE, Baron-Cohen S, Calder A, Keane J, Young A. Acquired theory of mind impairments in individuals with bilateral amygdala lesions. Neuropsychologia. 2003;41(2):209-20. doi: 10.1016/s0028-3932(02)00151-3. PMID 12459219
- [Derived] Yrondi A, Aouizerate B, El-Hage W, Moliere F, Thalamas C, Delcourt N, Sporer M, Taib S, Schmitt L, Arlicot N, Meligne D, Sommet A, Salabert AS, Guillaume S, Courtet P, Galtier F, Mariano-Goulart D, Champfleur NM, Bars EL, Desmidt T, Lemaire M, Camus V, Santiago-Ribeiro MJ, Cottier JP, Fernandez P, Meyer M, Dousset V, Doumy O, Delhaye D, Capuron L, Leboyer M, Haffen E, Peran P, Payoux P, Arbus C. Assessment of Translocator Protein Density, as Marker of Neuroinflammation, in Major Depressive Disorder: A Pilot, Multicenter, Comparative, Controlled, Brain PET Study (INFLADEP Study). Front Psychiatry. 2018 Jul 24;9:326. doi: 10.3389/fpsyt.2018.00326. eCollection 2018. PMID 30087626